CLINICAL TRIAL: NCT00237120
Title: Efficacy, Safety and Long-term Prognosis of Imatinib in Patients Newly Diagnosed With Chronic Myelogenous Leukemia (Chronic Phase)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571AJP02
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Myelogenous Leukemia in Chronic Phase
Keywords: Chronic Myelogenous Leukemia; Imatinib; CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib

SUMMARY:
This study will assess the safety and efficacy of imatinib in newly enrolled previously untreated patients with chronic phase CML.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Chronic Myelogenous Leukemia in Chronic Phase
* Previously untreated with Interferon-alpha
* Performance status is normal or capable of only limited self-care

Exclusion Criteria:

* Patients who are pregnant or possibly pregnant
* Significant hepatic diseases
* Chronic Myelogenous Leukemia in advanced phase

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 15 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2002-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
3 years overall survival
Duration of remaining in chronic phase

SECONDARY OUTCOMES:
Cytogenetic response and hematologyc response in every 3 or 6 months with 3 years treatment of Imatinib,
Adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis